CLINICAL TRIAL: NCT00997165
Title: Impact of Adipose Tissue Repartition on the Time Course of Vascular Dysfunction - the NUMEVOX Cohort
Acronym: NUMEVOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Pierre Henri Ducluzeau/MD-PhD, UH Angers
Other Study IDs: CHU-Promoteur 08-01
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Metabolic Diseases; Sleep Apnea; Atherosclerosis
Keywords: fatty liver; adipose tissue
MeSH Terms: conditions — Metabolic Diseases; Sleep Apnea Syndromes; Atherosclerosis; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Metabolic syndrome (MS): Patients suspected of metabolic syndrome without sleep apnea or liver steatosis
- MS with sleep apnea: Metabolic syndrome with sleep apnea
- MS with Liver steatosis: Metabolic syndrome with liver steatosis

SUMMARY:
The NUMEVOX cohort is intended to follow-up the macro and microvascular dysfunction in relation to adipose tissue repartition in patients with metabolic syndrome associated to liver steatosis, sleep apnea. Duration of the follow-up is 3 years for each patient entering the cohort.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age > 18 years old
* suspected of metabolic syndrome
* affiliated to french social health care

Exclusion Criteria:

* age < 18 years old
* pregnancy
* no informed consent
* not eligible for the study (no MS, cancer)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient suspected of metabolic syndrome with or without sleep apnea or liver steatosis.
  Informed consent with signature.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-03 (Estimated); Study Completion 2017-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: pierre henri Ducluzeau, MD PhD, Study Director — UH Angers
Locations (1):
- Pôle Maladies Métaboliques et Médecine Interne, Angers, France